CLINICAL TRIAL: NCT03471858
Title: MEchanical DIlatation of the Cervix in a Scarred Uterus (MEDICS)
Brief Title: Mechanical Dilation of the Cervix in a Scarred Uterus
Acronym: MEDICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Singapore (Other Government)
Collaborators: Department of Obstetrics and Gynaecology, National University Hospital (Unknown); Yong Loo Lin School of Medicine (Other); National University Hospital, Singapore (Other); National University of Singapore (Other)
Responsible Party: Principal Investigator, Soe-na Choo, Medical Officer, Ministry of Health, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/00248
Record Dates: First submitted 2018-03-13; First posted 2018-03-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Related; Labor Complication; Cesarean Section; Dehiscence
Keywords: caesarean, uterus
MeSH Terms: conditions — Obstetric Labor Complications | interventions — Prostaglandins; KLK15 protein, human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cervical Balloon (Active Comparator): Transcervical 2-way 18 French (18F) single balloon Foley catheter, applied using a sponge-holding forceps into the cervical canal with the balloon inflated to a minimum of 30ml and maximum of 60ml with sterile water or saline [1]. This will be administered once during the study and will be retained for a maximum of 12 hours within the 24 hour study period.
  Interventions: Device: Cervical balloon
- Prostaglandin (Active Comparator): Prostaglandin E2 (Prostin®) 3mg tablet, placed high in the vaginal fornix. This will be administered per vaginum once in the first 6 hours; a second dose is administered at the discretion of the clinician / clinical team 6 hours after the first pessary, for a cumulative total of 6mg within the 24 hour study period.
  Interventions: Drug: Prostaglandins

INTERVENTIONS:
Device: Cervical balloon — To assess if a cervical balloon catheter (foleys catheter) for mechanical induction of labour is comparable to prostaglandin usage for induction of labour in women who have had a previous caesarean section.
  Other Names: Foley Balloon Catheter
  Arms: Cervical Balloon
Drug: Prostaglandins — Prostin will be used in the control arm.
  Other Names: Prostin
  Arms: Prostaglandin

SUMMARY:
To determine if mechanical labour induction can offer a safer and effective alternative to prostaglandins to women with previous caesarean section attempting trial of labour after caesarean (TOLAC).

DETAILED DESCRIPTION:
There is good evidence to show that induction of labour with a transcervical balloon compares favourably with the use of prostaglandins.The cervical balloon works by softening & stretching the cervix mechanically & stimulates the release of endogenous prostaglandins.

When compared with prostaglandins, meta-analysis have shown that for TCB induction, there is no significant different in caesarean section rates (27% vs 25%) with a reduced risk of hyperstimulation with fetal heart rate change (0.4% vs 3%). Further, when compared against induction with misoprostol, induction with a Foley catheter balloon was found to have a lower rate of caesarean section for a non-reassuring fetal heart rate (RR 0.54, 95% CI 0.37-0.79) and a fewer vaginal instrumental deliveries (RR 0.74, 95% CI 0.55-0.95) [41]. One randomized controlled trial of 824 women with no previous caesarean section comparing foley catheter balloon with a prostaglandin E2 gel demonstrated no difference in caesarean section rates & 2 cases of uterine rupture or perforation in the prostaglandin E2 arm but not in the foley catheter balloon arm. Another study involving 1859 women comparing foley catheter balloon with oral misoprostol showed no difference in caesarean section rates or complications. It was, however, noted that induction with foley catheter balloon more likely required oxytocin induction at 80.3% vs 68.4% for misoprostol.

While there were earlier concerns of an increase in infectious morbidity when using mechanical induction of labour due to the presence of a foreign body, more recent RCTs & meta-analysis have shown that there is no significant increase.

One of the main concerns for induction of labour in patients with a previous uterine scar is an increased risk of uterine rupture. One observational study of 20,095 women quoted a risk of uterine rupture in spontaneous labour to be 0.52% & in prostaglandin-induced labour to be 0.77%. Another observational study involving 33,699 women quoted a risk of 0.4% and 1% respectively. While there are also studies which suggest that there is no significant increase in the rate of uterine rupture, many professional bodies have discouraged prostaglandin-induction in women with previous scars.

Due to lower levels of hyperstimulation that could lead to fetal distress or uterine rupture, trans cervical balloon induction has found itself as a possible, safer means of induction of labour for women who are keen for vaginal birth after caesarean and are agreeable with induction. Most RCTs were small in size & did not demonstrate any uterine rupture or dehiscence. However, 2 retrospective cohort studies involving a size of 2479 & 208 women respectively showed a uterine rupture rate of about 0.5%. trans cervical balloon induction appears to be a safe method for inducing consenting women keen for vaginal birth after caesarean and this study will contribute towards this body of evidence.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 21 years of age at booking visit
* 1 previous uncomplicated lower segment caesarean section (CS)
* Aiming for TOLAC
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study
* Singleton pregnancy
* Gestational age >37 weeks
* Understands risk of TOLAC
* Eligible for induction of labour for the standard obstetric indications, including post-date or post-term pregnancies at 40-41 completed weeks of gestation
* Unfavourable Bishop's Score ≤ 5 requiring cervical priming
* Previous uterine surgery, including simple myomectomy, where there is no contraindication to TOLAC
* Reactive CTG pre-induction
* Ruptured membranes

Exclusion Criteria:

* Refusal to participate
* Women with 2 or more previous CS
* Previous classical or lower segment vertical incision, or inverted T or J incision in the previous caesarean delivery
* Previous uterine surgery with contra-indication to future TOLAC
* Maternal contraindication for vaginal delivery
* Fetal contraindication for vaginal delivery or major fetal abnormality
* Malpresentation or cord presentation
* Placenta praevia <20mm from internal os
* Chorioamnionitis
* Antepartum haemorrhage of undetermined origin AND deemed a contraindication for TOLAC
* Suspected fetal macrosomia (estimated weight on ultrasound >4kg) AND deemed a contraindication for TOLAC
* Congenital uterine abnormality
* Multifetal pregnancy
* Latex allergy or poorly-controlled asthma

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant females
Enrollment: 44 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2022-08-27 (Actual); Study Completion 2025-08-16 (Actual)

PRIMARY OUTCOMES:
Improvement in Bishops score | 24hours
  Assess for increase in Bishops score from baseline of <5 (Unfavourable) to >6

SECONDARY OUTCOMES:
Achieving active labour | Within 24-48hours of intervention
  Achieving delivery
Number of PGE tablets required | Within 24-48hours of intervention
  For the prostin arm - How many tablets required, ie 1 or 2 to achieve improvement in Bishops score
Number of times the foley catheter (cervical balloon) needs to be readjusted | Within 24-48hours of intervention
  Numerical number of the times the foley catheter needs to be removed, replaced or readjusted
Mode of delivery | Within 24-48hours of intervention
  Successful vaginal birth after previous caesarean section, or emergency caesarean section
Maternal complications | Within 24-48hours of intervention
  failed device insertion, inability to void urine following insertion, intolerance of device and early removal, vaginal bleeding after insertion of device, spontaneous membrane rupture.
Fetal complications | Within 24-48hours of intervention
  fetal distress, meconium-stained liquor, malpresentation, neonatal Apgar score of <7 at 5 minutes, cord blood pH of ≤7.0, admission to NICU, neonatal hypoxic-ischaemic encephalopathy, neonatal death.
Infectious complications | Within 24-48hours of intervention
  intrauterine infection, maternal sepsis (e.g. endometritis, UTI), neonatal sepsis, maternal pyrexia, onset of antibiotics
Labour complications | Within 24-48hours of intervention
  uterine hyperstimulation (i.e. >5 contractions / 10mins with abnormal CTG), placental abruption, cord prolapse, postpartum haemorrhage, 3rd / 4th degree perineal tears, uterine rupture.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choo SN, Kanneganti A, Abdul Aziz MNDB, Loh L, Hargreaves C, Gopal V, Biswas A, Chan YH, Ismail IS, Chi C, Mattar C. MEchanical DIlatation of the Cervix-- in a Scarred uterus (MEDICS): the study protocol of a randomised controlled trial comparing a single cervical catheter balloon and prostaglandin PGE2 for cervical ripening and labour induction following caesarean delivery. BMJ Open. 2019 Nov 6;9(11):e028896. doi: 10.1136/bmjopen-2019-028896. PMID 31699720